CLINICAL TRIAL: NCT07115290
Title: Comparative Evaluation of Glass Ionomer and Resin-Based Fissure Sealants on Newly Erupted Permanent First Molars: A 24-Month Randomized Clinical Trial
Acronym: FISSURE24
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulcin Bulut (Other)
Responsible Party: Sponsor-Investigator, Gulcin Bulut, Associate Professor, DDS, PhD, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 612-SBKAEK; TİTCK-2023-067 (Other: Turkish Medicines and Medical Devices Agency)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries; Fissure Sealants; Permanent Molars; Child; Healthy Volunteers
Keywords: Dental caries; Fissure sealant; Glass ionomer; Resin-based sealant; Moisture-tolerant; Retention; Permanent molar; Children; Split-mouth design; Randomized clinical trial; Marginal adaptation; USPHS criteria
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: This study employed a split-mouth crossover design in which each participant received both interventions. One first permanent molar on the right or left side of the same dental arch was sealed with a glass ionomer-based sealant, while the contralateral molar on the opposite side of the same arch received a moisture-tolerant resin-based sealant. This design minimizes inter-subject variability and allows for a direct comparison within the same oral environment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glass Ionomer Sealant Arm (Active Comparator): In this arm, a high-viscosity glass ionomer-based fissure sealant (Fuji Triage™ Capsule, GC Corporation, Tokyo, Japan) was applied to one of the newly erupted permanent first molars of each participant using a split-mouth design.
  Interventions: Device: Glass ionomer-based fissure sealant
- Resin-Based Sealant Arm (Active Comparator): In this arm, a moisture-tolerant resin-based fissure sealant (UltraSeal XT® Hydro, Ultradent Products Inc., South Jordan, UT, USA) was applied to the contralateral newly erupted permanent first molar of the same participant, using the split-mouth method.
  Interventions: Device: Resin-based fissure sealant

INTERVENTIONS:
Device: Glass ionomer-based fissure sealant — A high-viscosity, self-curing glass ionomer sealant used for the occlusal surfaces of newly erupted permanent molars. This material releases fluoride and is moisture-tolerant during application. The product used in this study was Fuji Triage™ Capsule (GC Corporation, Japan).
  Other Names: Fuji Triage; Glass ionomer fissure sealant; GC Fuji Triage; GIC sealant
  Arms: Glass Ionomer Sealant Arm
Device: Resin-based fissure sealant — A moisture-tolerant, light-cured resin-based fissure sealant designed for application to occlusal surfaces in partially erupted permanent molars. The material exhibits strong adhesion in moist conditions and forms a durable barrier against caries. The product used in this study was UltraSeal XT® Hydro (Ultradent Products Inc., USA).
  Other Names: UltraSeal XT Hydro; Moisture-tolerant resin sealant; Hydrophilic sealant
  Arms: Resin-Based Sealant Arm

SUMMARY:
This clinical study aims to compare the clinical performance of two different fissure sealant materials-glass ionomer and resin-based-when applied to newly erupted permanent first molars in children. The study evaluates which material provides better retention, marginal adaptation, and protection against dental caries over a 24-month period.

DETAILED DESCRIPTION:
This randomized, split-mouth, clinical study was designed to compare the clinical effectiveness of two different fissure sealant materials-glass ionomer-based (Fuji Triage™ Capsule) and moisture-tolerant resin-based (UltraSeal XT® Hydro)-in newly erupted permanent first molars in children aged 6-7 years.

The study evaluates the retention rates, marginal adaptation, marginal discoloration, and the ability of each material to prevent dental caries over a 24-month follow-up period. A total of 70 teeth from 35 children were sealed using a split-mouth design, ensuring that each participant received both types of sealants on contralateral molars. Clinical evaluations were performed at 1, 6, 12, 18, and 24 months using modified United States Public Health Service (USPHS) criteria.

The goal of the study is to determine whether the moisture-tolerant resin-based material offers a clinical advantage in terms of sealant retention and caries prevention in a partially erupted, moisture-challenged clinical environment.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-7 years
* Children who are systemically healthy and classified as ASA I and II16
* Children whose parents and themselves have agreed to attend the study and follow-up visits throughout the study period
* Children who have established oral hygiene habits

Exclusion Criteria:

* Children whose caregivers did not sign the informed consent form, and patients who wished to withdraw or for whom the treatment protocol was not properly followed.
* Children who have restorations, cavitated surfaces or developmental defects and hypoplasia on the permanent first molar teeth to be treated.
* Medically compromised and children who need special treatment.
* History of adverse reactions to any restorative materials.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Sealant retention | 1, 6, 12, 18, and 24 months
  Assessment of the retention of the fissure sealant material on the occlusal surface of the first permanent molars using modified USPHS criteria. Evaluated at 1, 6, 12, 18, and 24 months.

SECONDARY OUTCOMES:
Marginal adaptation | 1, 6, 12, 18, and 24 months
  Evaluation of the marginal adaptation of the sealant to the tooth structure using modified USPHS criteria.
Marginal discoloration | 1, 6, 12, 18, and 24 months
  Assessment of any marginal discoloration of the sealant using modified USPHS criteria.
Presence of caries | 1, 6, 12, 18, and 24 months
  Detection of carious lesions on sealed occlusal surfaces throughout the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Gulcin F Bulut, DDS, PhD, Principal Investigator — Dokuz Eylul University, Faculty of Dentistry, Department of Pediatric Dentistry
Locations (1):
- Dokuz Eylul University, Faculty of Dentistry, Department of Pediatric Dentistry, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No